CLINICAL TRIAL: NCT02578810
Title: Sensitivity and Specificity of Bispectral Index (BIS) EEG Parameter, sFIT (Soluble FMS Tyrosine Kinase): PIGF (Placental Growth Factor) Ratio, Adrenomedullin for Grading Preeclampsia Integrated Estimate Risk Score (PIERS)
Brief Title: PIERS and BIS, sFIT:PIGF, Adrenomedullin
Acronym: BIS2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Suez Canal University (Other)
Collaborators: University of Malaya (Other)
Responsible Party: Principal Investigator, Ashraf A. Dahaba, Principle Investigator, Suez Canal University
Other Study IDs: MUGraz2
Record Dates: First submitted 2015-10-15; First posted 2015-10-19 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Eclampsia
MeSH Terms: conditions — Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Eclampsia: In 24 patients with Eclampsia or pre-eclampsia investigators will use an artefact-free 20-min mean BIS value, as well as biomarkers sFIT (soluble FMS-like Tyrosine Kinase): PIGF (Placental Growth Factor) ratio and adrenomedullin mortality risk stratifier to classify the degree of pre-eclampsia correlated the PIERS Pre-eclampsia risk assessment PIERS percentage (http://piers.cfri.ca/PIERSCalculatorH.aspx) will be calculated from patients' clinical and laboratory findings documented in their charts.
- Control: In 24 control patients without Eclampsia or pre-eclampsia investigators will use an artefact-free 20-min mean BIS value, as well as biomarkers sFIT (soluble FMS-like Tyrosine Kinase): PIGF (Placental Growth Factor) ratio and adrenomedullin mortality risk stratifier to classify the degree of pre-eclampsia correlated the PIERS Pre-eclampsia risk assessment PIERS percentage (http://piers.cfri.ca/PIERSCalculatorH.aspx) will be calculated from patients' clinical and laboratory findings documented in their charts

SUMMARY:
Pre-eclampsia, more than being proteinuric gestational hypertension alone, is a state of exaggerated systemic inflammation and remains a leading direct cause of maternal morbidity and mortality worldwide.1 Standardization of antenatal and postnatal assessment and surveillance of pre-eclampsia with protocols that recognize the systemic inflammatory model of preeclampsia have been associated with reduced maternal morbidity.

DETAILED DESCRIPTION:
Background: Pre-eclampsia, more than being proteinuric gestational hypertension alone, is a state of exaggerated systemic inflammation and remains a leading direct cause of maternal morbidity and mortality worldwide.1 Standardization of antenatal and postnatal assessment and surveillance of pre-eclampsia with protocols that recognize the systemic inflammatory model of preeclampsia have been associated with reduced maternal morbidity.2 To quantitatively asses electroencephalography (EEG) mental involvement in Pre-eclampsia is still time consuming and not always readily available. PIERS was developed and internally validate as a pre-eclampsia outcome prediction model- (Preeclampsia Integrated Estimate of RiSk) model.3 The purpose of our study was to evaluate the discriminative power of the Bispectral Index (BIS), biomarkers sFIT (soluble FMS-like Tyrosine Kinase): PIGF (Placental Growth Factor) ratio,4 and adrenomedullin mortality risk stratifier,5 to classify the degree and progression of pre-eclampsia.

Methods: In 24 patients with Eclampsia or pre-eclampsia investigators will use an artefact-free 20-min mean BIS value, as well as biomarkers sFIT (soluble FMS-like Tyrosine Kinase): PIGF (Placental Growth Factor) ratio and adrenomedullin mortality risk stratifier to classify the degree of pre-eclampsia correlated the PIERS Pre-eclampsia risk assessment PIERS percentage (http://piers.cfri.ca/PIERSCalculatorH.aspx) will be calculated from patients' clinical and laboratory findings documented in their charts, compared with 24 pregnant patients without Eclampsia or pre-eclampsia.

ELIGIBILITY:
Inclusion Criteria

1. Pregnancy at any stage (3 trimesters)
2. Eclampsia (Frank eclampsia) will be the crux of the study
3. Pre-eclampsia that is suspected will end up with Frank Eclampsia

Exclusion criteria:

1. Any neurological conditions that can alter the electroencephalography like epilepsy
2. Any medical conditions that can alter the electroencephalography like hypoglycemia

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 24 patients with Eclampsia or pre-eclampsia investigators will use an artefact-free 20-min mean BIS value, as well as biomarkers sFIT (soluble FMS-like Tyrosine Kinase): PIGF (Placental Growth Factor) ratio and adrenomedullin mortality risk stratifier to classify the degree of pre-eclampsia correlated the PIERS Pre-eclampsia risk assessment PIERS percentage (http://piers.cfri.ca/PIERSCalculatorH.aspx) will be calculated from patients' clinical and laboratory findings documented in their charts, compared with 24 pregnant patients without Eclampsia or pre-eclampsia
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2016-10; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Decline in BIS | we will record Bispectral Index (BIS) for a quite 20 min no tactile contact or noise that could raise the BIS inadvertently
  our hypothesis is that a decline of Bispectral Index (BIS) assuming to be in the range of 15-60 will correlate to the with a high PIERS we can then quantify this BIS decline maybe in 4 Eclampsia grades

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Dahaba, MD, Principal Investigator — Guest Professor
Locations (1):
- Medical Ethics Committee, University Malaya Medical Centre, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No